CLINICAL TRIAL: NCT00358345
Title: PHP Preferential Hyperacuity Perimeter for the Detection of Choroidal Neovascularization
Brief Title: PreView PHP Preferential Hyperacuity Perimeter for the Detection of Choroidal Neovascularization
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Osnat Ehrman, NotalVision
Organization: Notal Vision Inc. (Industry)
Other Study IDs: PHP C9
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Intermediate AMD
- 2: Newly diagnosed CNV

SUMMARY:
The primary objective of this study is to assess the ability of the PreView PHP(study device)to detect newly diagnosed non-treated Choroidal Neovascularization (CNV)lesion associate with advanced Age-related Macular Degeneration (AMD) or Myopia and differentiate them from Intermediate AMD or Geographic Atrophy (GA)or patients with high Myopia with no CNV.

This study secondary is to enhance NotalVision normative database.

DETAILED DESCRIPTION:
* The study is prospective, multi-center, comparative study.
* A clinical trail with FDA approval device (510K).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (up yo 2 months) CNV OR Intermediate AMD
* Age >50 for AMD subjects
* Age >18 for Myopic subjects
* VA 20/160 or better in the study eye
* Mental and physical ability to performed a PHP test

Exclusion Criteria:

* Evidence of macular disease other than AMD or high myopia in the study eye.
* Previous surgical or laser treatment within the macular erea.
* Concurrent intraocular drug therapy (within 30 days).
* Present of any significant media opacity that preclude a clear veiw of the macula.
* Any non macular related ocular surgery performed within 3 months prior to the study.
* CNV subjects inability to tolerate intravenous fluorscien angiography.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 200 subjects with intermediate AMD in at least one (1) eye based on medical record review and/or clinical diagnosis and at least 200 subjects with neovascular AMD in at least one (1) eye.
Sampling Method: Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2003-10; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Sharon, MD, Study Director — Notal Vision
Locations (1):
- Tel Aviv Sourasky medical center, Tel Aviv, Israel